CLINICAL TRIAL: NCT06969079
Title: Effectiveness of Ba Duan Jin Exercise on Chronic Insomnia (CI) With Hyperarousal/Anxiety
Brief Title: Ba Duan Jin for CI With Hyperarousal/Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI+HA-BDJ
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Mind-Body Therapies; Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ba Duan Jin Exercise plus Sleep Hygiene Education (Experimental)
  Interventions: Behavioral: Ba Duan Jin Exercise plus Sleep Hygiene Education
- Sleep Hygiene Education Only (Active Comparator)
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Ba Duan Jin Exercise plus Sleep Hygiene Education — Participants will receive Ba Duan Jin exercise combined with Sleep Hygiene Education. The Ba Duan Jin intervention consists of eight traditional Chinese Qigong movements performed daily for 6 weeks, with each session lasting 50 minutes, accompanied by structured sleep hygiene counseling.
  Arms: Ba Duan Jin Exercise plus Sleep Hygiene Education
Behavioral: Sleep Hygiene Education — Participants will receive Sleep Hygiene Education (SHE) alone, consisting of guidance on establishing healthy sleep habits, optimizing sleep environment, adjusting sleep schedules, reducing stimulants (e.g., caffeine, alcohol), and minimizing sleep-disruptive behaviors.
  Arms: Sleep Hygiene Education Only

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of Ba Duan Jin exercise in treating chronic insomnia (CI) with comorbid hyperarousal and anxiety symptoms.

DETAILED DESCRIPTION:
Chronic Insomnia (CI) is a common sleep disorder characterized by persistent difficulties in initiating or maintaining sleep, leading to significant daytime dysfunction. Many CI patients experience hyperarousal, both physiological and psychological, commonly manifested as anxiety, which further exacerbates sleep disturbances and reduces quality of life.

While pharmacotherapy and cognitive behavioral therapy (CBT) are effective for some patients, they are limited by side effects, costs, and accessibility. Traditional mind-body practices such as Ba Duan Jin, a classic Chinese Qigong exercise, have been explored as alternative therapies to improve sleep quality and alleviate anxiety symptoms.

Ba Duan Jin consists of a sequence of gentle and flowing movements designed to promote physical and mental relaxation. Preliminary studies suggest that mind-body exercises like Ba Duan Jin can positively influence sleep patterns, psychological well-being, and overall health.

This randomized controlled trial will recruit 84 participants diagnosed with CI and comorbid hyperarousal/anxiety symptoms. Participants will be randomly assigned to either a Ba Duan Jin plus Sleep Hygiene Education (SHE) group or an SHE-only group.

The intervention will last for 6 weeks, with participants in the Ba Duan Jin group practicing once daily for 50 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Insomnia Disorder according to DSM-5 criteria.
2. Pittsburgh Sleep Quality Index (PSQI) total score > 5.
3. Age ≥ 8 years.
4. Educational level of at least junior high school.
5. Voluntarily agree to participate and sign informed consent.
6. Presence of anxiety symptoms, defined as a Hamilton Anxiety Rating Scale (HAMA-14) score ≥ 14.

Exclusion Criteria:

1. Presence of severe physical illnesses or major psychiatric disorders, or assessed to be at risk of suicide.
2. Diagnosis or suspicion of sleep breathing disorder, restless legs syndrome, circadian rhythm sleep disorder, or engaged in night-shift work.
3. Pregnancy or breastfeeding.
4. Currently undergoing any form of psychological therapy.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 6 weeks | Baseline, 6 weeks
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of PSQI total scores from baseline to 3 months, 6 months, and 12 months | Baseline, 3 months, 6 months, 12 months
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.
The change of Insomnia severity index (ISI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.
The change of Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The DBAS assessing sleep related cognitions in 16 items rated on a 10-point Likert scale, and the total score ranges from 0 to 160 with higher scores indicating more intensive dysfunctional beliefs.
The change of sleep efficiency from baseline to 6 weeks, 3 months, 6 months, and 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
Change from Baseline in Snaith-Hamilton Pleasure Scale (SHAPS) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
The change of Short Form 36 (SF-36) total scores from baseline to 6 weeks, 3 months, 6 months, 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The SF-36 quantifying the quality of life in relation to health status consists of 36-items with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The total score ranges from 0-100 (the worst possible to the most possible).
The change of Patient Health Questionnaire-4 (PHQ-4) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-4 comprises a 2-item depression scale and a 2-item anxiety scale. Each instrument can reach values from 0-6. Higher Scores are indicating higher distress.
The change of Beck Depression Inventory (BDI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BDI assessing the existence and severity of symptoms of depression consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms.
The change of Beck Anxiety Inventory (BAI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BAI assessing the existence and severity of symptoms of anxiety consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe anxiety.
The change of Patient Health Questionnaire-15 (PHQ-15) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-15 measuring somatic distress consists of 15 items, and the total score ranges from 0 to 30 with higher scores indicating more severe somatic distress
The change of 5-item Perceived Deficits Questionnaire-Depression (PDQ-D-5) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PDQ-D-5 assessing perceived cognitive deficits from the patient's perspective consists of 5 items, and the total score ranges from 0 to 20 with higher scores indicating greater perceived deficit.
The change of Life Events Scale (LES) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The LES assessing the perceived stress and number of stressful life events experienced consists of 48 items which are classified into three dimensions: family life events (28 items), work and study events (13 items), and social events (7 items) with higher scores in LES perceived greater stressfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan B, Song W, Zhang J, Er Y, Xie B, Zhang H, Liao Y, Wang C, Hu X, Mcintyre R, Lee Y. The efficacy of mind-body (Baduanjin) exercise on self-reported sleep quality and quality of life in elderly subjects with sleep disturbances: a randomized controlled trial. Sleep Breath. 2020 Jun;24(2):695-701. doi: 10.1007/s11325-019-01999-w. Epub 2020 Jan 2. PMID 31898191